CLINICAL TRIAL: NCT01824537
Title: Transmission Reduction and Prevention With HPV Vaccination (TRAP-HPV) Study: A Randomized Controlled Trial of the Efficacy of HPV Vaccination in Preventing Transmission of HPV Infection in Heterosexual Couples
Brief Title: Transmission Reduction and Prevention With HPV Vaccination (TRAP-HPV) Study
Acronym: TRAP-HPV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Eduardo Franco, James McGill Professor and Chair, Department of Oncology; Director, Division of Cancer Epidemiology, McGill University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIHR-MOP-125949; IIS #38265 (Other Grant/Funding Number: Merck); MOP-125949 (Other Grant/Funding Number: Canadian Institutes of Health Research); FDN-143347 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Human Papillomavirus Infection
Keywords: Human papillomavirus (HPV); Vaccination; Cervical cancer prevention; Herd immunity
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines; Human Papillomavirus Recombinant Vaccine nonavalent; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HPV vaccine, Gardasil 9 (Active Comparator): HPV vaccine intervention: The intervention vaccine will be Gardasil 9, a 9-valent vaccine by Merck. This vaccine was chosen because it allows for the observation of 9 HPV outcomes (HPV 6, 11, 16 and 18) (the other available vaccine, Cervarix, protects against HPVs 16 and 18, only).
  Interventions: Biological: HPV vaccine, Gardasil 9
- Hepatitis A vaccine (Placebo Comparator): The placebo comparator will be Avaxim, by Sanofi Pasteur. This control vaccine was chosen because hepatitis A immunization provides a similar health prevention incentive as HPV vaccination to study participants while preserving the scientific cogency of a "placebo" comparator. Gardasil 9 requires administration of 3 doses, while Avaxim only requires 2 doses. For this reason, a placebo injection (saline solution) will be added in between the Avaxim vaccination regimen. Consequently, both treatment and control vaccines will have similar regimens, i.e., study entry, 2 months, and 6 months.
  Interventions: Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: HPV vaccine, Gardasil 9 — Once recruited, both individuals in a couple will be randomized independently to Gardasil 9 or placebo (Avaxim).
  Arms: HPV vaccine, Gardasil 9
Biological: Hepatitis A vaccine — Provided by Sanofi Pasteur.
  Other Names: Avaxim
  Arms: Hepatitis A vaccine

SUMMARY:
Human papillomavirus (HPV) is a member of the Papillomaviridae family of DNA viruses that is capable of infecting humans. HPV infection can cause cancers of the cervix, vulva, vagina, and anus in women or cancers of the anus and penis in men. Two prophylactic vaccines have been proven to be highly effective in preventing the acquisition of HPV infection and the genital precancerous lesions caused by it. However, we do not know yet if a previously infected individual, once vaccinated, would be less infective to her or his sexual partner. We plan to conduct a study, called Transmission Reduction And Prevention with HPV vaccination (TRAP-HPV) study to answer this question. It will include 500 sexually active couples* (total of 1000 individuals) in university student health clinics in Montreal (age 18-45 years). It will be a randomized placebo-controlled, double-blinded intervention trial. Study participants will be followed up to 12 months. Behavioural and biological data will be collected at the time of study enrolment, then at months 2, 4, 6, 9 and 12 post-enrolment. The results of this trial will be invaluable in informing policies regarding vaccination of women and men.

DETAILED DESCRIPTION:
Two prophylactic vaccines (Gardasil by Merck, and Cervarix by GlaxoSmithKline) have been proven in randomized controlled trials (RCT) to be highly effective in preventing infection against the target HPV types (HPV-6, 11, 16 and 18, for Gardasil, and HPV-16/18, for Cervarix) and the cervical precancerous lesions caused by them. These vaccines have shifted the paradigm of prevention and are expected to have a major impact in reducing the burden of cervical cancer and of other HPV-associated malignancies, such as vulvar, vaginal, penile, anal, and oropharyngeal cancers, as well as benign HPV-associated conditions (in the case of Gardasil), such as anogenital warts and respiratory papillomatosis. However, little is known about the extent with which vaccination may reduce transmission between sexual partners; i.e. much remains to be understood on the effects of HPV vaccine in preventing transmission of target HPV types to sexual partners of vaccinated individuals and its impact on herd immunity.

The investigators propose to conduct a placebo-controlled, double-blinded RCT to measure the impact of vaccination in preventing HPV transmission within young (age 18-45) heterosexual couples at McGill and Concordia Universities in Montreal, Canada. Individual partners in 500 couples* will be randomized to a treatment (Gardasil 9) or a control vaccine (Avaxim, a hepatitis A vaccine). This control vaccine provides a similar health benefit incentive as HPV vaccination while preserving the scientific cogency of a "placebo" comparator. Risk factor data will be collected via computerized questionnaires at enrolment (time 0), 2, 4, 6, 9 and 12 months*. At all time points, the investigators will measure HPV DNA infection status by polymerase chain reaction (PCR) in both partners in exfoliated penile, and oral samples from men and vaginal, oral samples from women. Assessing pre-enrolment humoral immune response to HPV infection with a competitive Luminex immunoassay (CLIA) will be done in an enrolment blood sample from all study participants.

The primary outcome will be the reduction of HPV DNA positivity for the target HPV vaccine types (types 6, 11, 16 and 18) in multiple anatomic sites in Avaxim-treated sexual partners of participants who received Gardasil 9. The investigators hypothesize that HPV vaccination is effective in reducing the risk of HPV transmission to their sexual partners. They will use the Kaplan-Meier technique and logrank tests to compare the cumulative probability of HPV infection in sexual partners of vaccinated versus unvaccinated individuals against follow-up time, and Cox proportional hazards regression to estimate the effect of vaccination and other covariates on transmission of HPV to sexual partners. Statistical analyses will follow an intention-to-treat approach but additional regression models will examine the role of several candidate determinants in mediating transmission and the protective effects. Mixed-effects models will also be used to take advantage of the repeated measurements across visits, HPV types, and anatomical sites for the same subject.

In addition to the findings on protection to unvaccinated partners, it is expected that this study will provide valuable insights as to whether protection may exist for a vaccine recipient in preventing infection in an anatomical site in which a target type has not yet established infection. These findings will generate key parameter data to inform the extent of herd immunity in cost-effectiveness models of HPV vaccination. Such models are essential to arrive at rational science-driven policies of HPV vaccination in girls and boys in Canada.

As of March 13, 2020, study visits were temporarily suspended due to the COVID-19 pandemic. With university approval, study visits were resumed as of May 26, 2020. Precautionary measures were put in place to minimize the risks related to exposure to the coronavirus. This included minimizing the number of participants present at the study site, using COVID-19 screening questionnaires prior to the visit, wearing personal protective equipment, disinfecting hands and common areas, and maintaining safe distancing. Transportation (by Taxi or Uber) or parking fees were also paid for to ensure safe distancing while traveling to the study site. The interruption in study visits due to the COVID-19 pandemic led to slight alterations in the timing of vaccinations, which will be adjusted for in the final analyses as required.

*With the slow accrual rates exacerbated by the COVID-19 pandemic, it was estimated that the target sample would not be reached within a reasonable timeframe. Therefore, we completed the study with 188 couples, before reaching the original target of 500 couples (1000 participants) and the interim target of 250 couples (500 participants) in order to maintain the scientific value of the study. In addition, we proposed to make the fifth time point the final visit. This shortened follow-up duration affected only three couples. Such protocol amendments were approved by the Institutional Review Boards.

Published protocol is available at PMID: 32788190

ELIGIBILITY:
Inclusion Criteria:

* Couple must have been in a new relationship that started no more than six months prior to study entry
* Both partners plan on remaining in Montreal for at least 1 year
* Plan on having continued sexual contact with partner
* Be willing to comply with study procedures

Exclusion Criteria:

* Volunteers must not have been vaccinated against HPV-Gardasil-9 (both partners)
* Any history of cervical, penile, oral or anal cancers
* Being pregnant or plan on immediately becoming pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 372 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariam El-Zein, PhD, Study Director — McGill University
Locations (1):
- McGill University - Division of Cancer Epidemiology, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] MacCosham A, El-Zein M, Burchell AN, Tellier PP, Coutlee F, Franco EL; TRAP-HPV study group. Protection to Self and to One's Sexual Partner After Human Papillomavirus Vaccination: Preliminary Analysis From the Transmission Reduction And Prevention with HPV Vaccination Study. Sex Transm Dis. 2022 Jun 1;49(6):414-422. doi: 10.1097/OLQ.0000000000001620. Epub 2022 Mar 2. PMID 35235550
- [Derived] MacCosham A, El-Zein M, Burchell AN, Tellier PP, Coutlee F, Franco EL. Transmission reduction and prevention with HPV vaccination (TRAP-HPV) study protocol: a randomised controlled trial of the efficacy of HPV vaccination in preventing transmission of HPV infection in heterosexual couples. BMJ Open. 2020 Aug 11;10(8):e039383. doi: 10.1136/bmjopen-2020-039383. PMID 32788190

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPV Vaccine, Gardasil 9 | Hepatitis A Vaccine
Started | 190 | 182
Completed | 112 | 95
Not Completed | 78 | 87
Not completed — Lost to Follow-up | 78 | 87

BASELINE CHARACTERISTICS:
Population: The analysis population includes 82.8% of the enrolled participants, consisting of 154 couples who had i) at least one follow-up visit, and ii) valid baseline genital samples from both partners, or imputation was possible based on subsequent visits in case a baseline genital sample was invalid. Participants (11 males and 9 females) received Gardasil up until July 8, 2015, after which they received Gardasil 9 (64 males and 74 females).
Groups:
- Female: Hepatitis A Vaccine; Male: Hepatitis A Vaccine: The placebo comparator will be Avaxim, by Sanofi Pasteur. This control vaccine was chosen because hepatitis A immunization provides a similar health prevention incentive as HPV vaccination to study participants while preserving the scientific cogency of a "placebo" comparator. Gardasil 9 requires administration of 3 doses, while Avaxim only requires 2 doses. For this reason, a placebo injection (saline solution) will be added in between the Avaxim vaccination regimen. Consequently, both treatment and control vaccines will have similar regimens, i.e., study entry, 2 months, and 6 months.
  Hepatitis A vaccine: Provided by Sanofi Pasteur.
- Female: HPV Vaccine, Gardasil 9; Male: HPV Vaccine, Gardasil 9: HPV vaccine intervention: The intervention vaccine will be Gardasil 9, a 9-valent vaccine by Merck. This vaccine was chosen because it allows for the observation of 9 HPV outcomes (HPV 6, 11, 16 and 18) (the other available vaccine, Cervarix, protects against HPVs 16 and 18, only).
  HPV vaccine, Gardasil 9: Once recruited, both individuals in a couple will be randomized independently to Gardasil 9 or placebo (Avaxim).
- Total: Total of all reporting groups
Arm/Group | Female: Hepatitis A Vaccine | Female: HPV Vaccine, Gardasil 9 | Male: Hepatitis A Vaccine | Male: HPV Vaccine, Gardasil 9 | Total
Number analyzed (Participants) | 71 | 83 | 79 | 75 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.2 (4.7) | 25.4 (6.2) | 25.7 (5.7) | 26.7 (6.9) | 25.5 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 83 | 0 | 0 | 154
  Male | 0 | 0 | 79 | 75 | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Birth Country: Canada | 39 | 41 | 36 | 36 | 152
  Birth Country: United States | 5 | 7 | 7 | 4 | 23
  Birth Country: Other: Brazil, China, Mexico, MENA, Sub-Saharan Africa, Latin America, Europe, Asia, Oceania | 27 | 34 | 36 | 35 | 132
  Birth Country: Missing | 0 | 1 | 0 | 0 | 1
Education [Count of Participants; unit: Participants]
  High school | 10 | 11 | 12 | 21 | 54
  College or vocational training | 10 | 15 | 16 | 14 | 55
  University | 51 | 57 | 50 | 40 | 198
  Missing | 0 | 0 | 1 | 0 | 1
Smoking Status [Count of Participants; unit: Participants] — A smoking status of "Former" includes participants who reported not being current smokers but reported smoking regularly in the past and/or reported having smoked at least 100 cigarettes in their lifetime.
  Participants
    Never | 52 | 60 | 59 | 45 | 216
    Former | 13 | 16 | 16 | 21 | 66
    Current | 6 | 6 | 3 | 9 | 24
    Missing | 0 | 1 | 1 | 0 | 2
Concurrent sex partners [Count of Participants; unit: Participants] — Any concurrent partners since the beginning of the relationship with TRAP-HPV partner, as reported at baseline.
  Participants
    No | 58 | 67 | 74 | 60 | 259
    Yes | 13 | 15 | 5 | 14 | 47
    Missing | 0 | 1 | 0 | 1 | 2
Number of lifetime vaginal sex partners [Median (Inter-Quartile Range); unit: partners] | 5 [2 to 14] | 6 [2 to 20] | 8 [3 to 15] | 7 [3 to 16] | 6 [2 to 15]
Age at coitarche [Median (Inter-Quartile Range); unit: years] | 17 [16 to 19] | 17.5 [16 to 19] | 18 [16 to 20] | 18 [16 to 19] | 18 [16 to 19]
Years since onset of sexual activity [Median (Inter-Quartile Range); unit: years] — Age at baseline minus age at coitarche.
  years | 4.8 [2.5 to 9.4] | 5.4 [2.5 to 9.8] | 6 [2.9 to 10.3] | 7.6 [3.1 to 12.6] | 5.8 [2.7 to 10.5]
Grouped HPV positivity [Count of Participants; unit: Participants] — Vaccine-targeted types include any of HPVs 6, 11, 16, 18, 31, 33, 45, 52, and 58.
  Any HPV includes any of 36 HPV types that were tested for: HPVs 6, 11, 16, 18, 26, 31, 33, 34, 35, 39, 40, 42, 44, 45, 51, 52, 53, 54, 56, 58, 59, 61, 62, 66, 67, 68, 69, 70, 71, 72, 73, 81, 82, 83, 84, and 89.
  Participants
    Vaccine-targeted (any 9vHPV) | 13 | 16 | 14 | 12 | 55
    Any HPV | 34 | 37 | 30 | 33 | 134

OUTCOME MEASURES:

1. Primary Outcome: HPV Incidence Rates, Expressed as Incident Infections/1000 Infection-months at Risk. These Were Calculated Separately for Females and Males Across the Four Vaccine Assignment Groups.
Description: Participants (n=308) from new (≤6 months) heterosexual couples aged 18+ in Montreal, Canada, were randomized into 4 groups:
  Group 1: 40 males and 40 females; Group 2: 31 males and 31 females; Group 3: 39 males and 39 females; Group 4: 44 males and 44 females. Genital samples, collected at 0, 2, 4, 6, 9, and 12 months, were genotyped for 36 HPV types. For females and males separately within each of the 4 groups, we calculated, via time-to-event analyses, the incidence rates (and their jackknife 95% confidence intervals, CI) as the number of incident infections/1000 infection-months at risk. We used type-specific HPV infections as the unit of analysis; that is, each participant could contribute time at risk for up to the 9 vaccine-targeted (i.e., HPVs 6, 11, 16, 18, 31, 33, 45, 52, and 58) type-specific HPV-level infections. Participants contributed time at risk for incidence of type-specific HPV-level infections if they had not previously tested positive for that HPV type.
Time Frame: Up to 12 months
Population: The analytical population consists of 82.8% of participants (154 couples=308 participants) who had at least one follow-up visit, and valid baseline genital samples from both partners or values imputed based on subsequent visits. Each participant contributed 9 observations, 1 for each of the 9 HPV types. In group 1, 720 units analyzed=80 participantsx9 HPV types. For each of the 4 groups, we report one incidence rate for males, and one for females, for a total of 8 incidence rate values.
Measure: Number (95% Confidence Interval); unit: incident infections/1000 infection-month
Units Other Than Participants: type-specific HPV (participant-HPV unit)
Groups:
- Group 1 - Male and Female: Hepatitis A Vaccine: Both participants of the couple were administered the active control Avaxim Hepatitis A vaccine, by Sanofi Pasteur. Gardasil 9 requires administration of 3 doses, while Avaxim only requires 2 doses. For this reason, a placebo injection (saline solution) was added in between the Avaxim vaccination regimen. Consequently, this regimen was given at study entry, 2 months, and 6 months.
- Group 2 - Male: Gardasil 9; Female: Hepatitis A Vaccine: The male was administered the Gardasil 9 vaccine, by Merck, while the female was administered the Avaxim Hepatitis A vaccine, by Sanofi Pasteur, with a placebo injection (saline solution) added in between the Avaxim vaccination regimen. Consequently, both treatment and active control vaccines had similar regimens, i.e., study entry, 2 months, and 6 months.
- Group 3 - Male: Hepatitis A Vaccine; Female: Gardasil 9: The male was administered the Avaxim Hepatitis A vaccine, by Sanofi Pasteur, with a placebo injection (saline solution) added in between the Avaxim vaccination regimen, while the female was administered the Gardasil 9 vaccine, by Merck. Consequently, both treatment and active control vaccines had similar regimens, i.e., study entry, 2 months, and 6 months.
- Group 4 - Male and Female: Gardasil 9: Both participants of the couple were administered the Gardasil 9 vaccine, by Merck. Gardasil 9 requires administration of 3 doses, which was given at study entry, 2 months, and 6 months.
Arm/Group | Group 1 - Male and Female: Hepatitis A Vaccine | Group 2 - Male: Gardasil 9; Female: Hepatitis A Vaccine | Group 3 - Male: Hepatitis A Vaccine; Female: Gardasil 9 | Group 4 - Male and Female: Gardasil 9
Number analyzed (Participants) | 80 | 62 | 78 | 88
Number analyzed (type-specific HPV (participant-HPV unit)) | 720 | 558 | 702 | 792
incident infections/1000 infection-month
  Female-HPV incidence rate: number analyzed (Participants) | 40 | 31 | 39 | 44
  Female-HPV incidence rate: number analyzed (type-specific HPV (participant-HPV unit)) | 360 | 279 | 351 | 396
  Female-HPV incidence rate | 1.40 [0.51 to 5.34] | 1.58 [0.55 to 6.17] | 1.05 [0.42 to 3.45] | 1.58 [0.71 to 4.25]
  Male-HPV incidence rate: number analyzed (Participants) | 40 | 31 | 39 | 44
  Male-HPV incidence rate: number analyzed (type-specific HPV (participant-HPV unit)) | 360 | 279 | 351 | 396
  Male-HPV incidence rate | 2.42 [0.97 to 7.63] | 0.99 [0.17 to 3.07] | 3.35 [1.95 to 6.30] | 1.67 [0.75 to 3.51]

ADVERSE EVENTS:
Time Frame: During the 12 months of follow up.
Description: Gardasil 9 and Avaxim are safe and approved vaccines, and the collection of oral and genital specimens for HPV testing are safe procedures. However, participants were prompted to contact the research nurse if they experienced any unusual or severe side effects throughout follow up.
Arm/Group | HPV Vaccine, Gardasil 9 | Hepatitis A Vaccine
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/182
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/182
Other Adverse Events (participants affected / at risk) | 0/190 | 0/182

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT01824537/Prot_SAP_000.pdf